CLINICAL TRIAL: NCT03644719
Title: Effectiveness of a Brief Cognitive and Behavioral Skills Program on Stage Transitions for Chronic Ketamine Abusers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University (Other)
Responsible Party: Principal Investigator, Tony Szu-Hsien Lee, Professor, National Taiwan University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Chronic Ketamine Abusers
Record Dates: First submitted 2018-08-12; First posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Substance Use Disorders
Keywords: Substance Abuse; Cognitive behavioral treatment; Ketamine; Stage of Change
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Two arms were used to examine the relative effect of the cognitive behavioral skills training (CBSR) and a time slot for education as usual (EAU). The CBST consists of six sessions. The first session is intended to establish rapport, build therapeutic cohesion through ice-breaking activities, and educate participants about the drug regulations stated in the Statute for Drug Hazard Prevention and Control. The following four sessions are devoted to interactively practicing refusal skills, communication skills, decision-making skills, and positive conflict resolution skills. The final session is to review what has been learned and reminds participants about the association of drug use with HIV/HCV.
Who Masked: Participant
Masking Description: Participants signed up for a time slot for cognitive behavioral skills training (CBST) or a time slot for education as usual (EAU), without being informed which was which.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavior skills training (Experimental): The first session is intended to establish rapport, build therapeutic cohesion through ice-breaking activities, and educate participants about the drug regulations stated in the Statute for Drug Hazard Prevention and Control. The following four sessions are devoted to interactively practicing refusal skills, communication skills, decision-making skills, and positive conflict resolution skills. The final session is to review what has been learned and reminds participants about the association of drug use with HIV/HCV.
  Interventions: Behavioral: Cognitive behavioral skills training
- Education as usual (No Intervention): The EAU group received six hours of informational lectures about ketamine, its effects on the brain, relevant regulations and laws, and the risks and modes of transmission of infectious diseases, including HIV and hepatitis C.

INTERVENTIONS:
Behavioral: Cognitive behavioral skills training — A brief cognitive behavioral skills training was applied to teach ketamine abusers about stimulus control, refusal skills, communication skills, decisional balance, and infectious diseases prevention.
  Arms: Cognitive behavior skills training

SUMMARY:
In recent years ketamine abuse becomes prevalent in youth in some Asian countries. Chronic ketamine abuse may lead to uropathology and cognitive impairments. No pharmacological interventions have been identified as effective for treating ketamine abuse or helpful in achieving or maintaining abstinence from ketamine. Cognitive-behavioral treatment is currently an important psychosocial intervention for addictive problems. This study aimed to test whether a brief cognitive-behavioral training program has a positive influence on stage transitions among ketamine abusers.

DETAILED DESCRIPTION:
409 ketamine abusers were recruited in this study, with 285 ketamine abusers participated in a 6-hour brief cognitive-behavioral intervention and 124 ketamine abusers attended educational lectures on ketamine abuse. A brief cognitive-behavioral intervention was applied to teach ketamine abusers about stimulus control, refusal skills, communication skills, decisional balance, and infectious diseases prevention. Stage of Change and knowledge about ketamine were assessed before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* ketamine use in 30 days
* more than 18 years old

Exclusion Criteria:

* no brain damage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2014-08-19 (Actual); Primary Completion 2017-03-19 (Actual); Study Completion 2017-03-19 (Actual)

PRIMARY OUTCOMES:
Motivation to change | 15 minutes
  Stage of Change Scale: Have you thought of abstaining from Ketamine? In 30 days? In six months?

SECONDARY OUTCOMES:
Knowledge about ketamine | 3 minutes
  5 items questionnaire about consequences of using ketamine: micturition, perception distortion, depression, behavioral inhibition and memory

CONTACTS AND LOCATIONS:
Overall Officials: Tony Szu-Hsien Lee, Ph.D., Principal Investigator — Health Promotion and Health Education

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baker A, Lee NK, Claire M, Lewin TJ, Grant T, Pohlman S, Saunders JB, Kay-Lambkin F, Constable P, Jenner L, Carr VJ. Brief cognitive behavioural interventions for regular amphetamine users: a step in the right direction. Addiction. 2005 Mar;100(3):367-78. doi: 10.1111/j.1360-0443.2005.01002.x. PMID 15733250
- See also: This study demonstrated that brief interventions consisting of cognitive behavior therapy increased the likelihood of abstinence from amphetamines among those receiving two or more treatment sessions. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Brief+cognitive+behavioural+interventions+for+regular+amphetamine+users%3A+a+step+in+the+right+direction.+Addiction